CLINICAL TRIAL: NCT05140772
Title: Evaluations the Effect of Parenteral Glutamine on Reducing Infection Morbidity in Burn Patients in ICU. A Randomized Controlled Double-blind Study.
Brief Title: Glutamine Effects in Burn Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, ashraf magdy eskandr, assistant professor of anesthesia, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19/5/2019 ANET4
Record Dates: First submitted 2021-10-19; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Drug Effect
MeSH Terms: interventions — alanylglutamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Active Comparator): Patient were received 0.5gm/kg/day IV glutamine infusion (dipeptiven 100ml contains 20 g N(2)-L-alanyl-L-glutamine (= 8.20 g L-alanine, 13.46 g L-glutamine) Water for Injections).
  Interventions: Drug: Dipeptiven
- group II (Placebo Comparator): Patients received an equivalent volume of normal saline daily for 7 days.
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: Dipeptiven — IV administration daily for 7 days
  Arms: group I
Drug: normal Saline — IV administration daily for 7 days
  Arms: group II

SUMMARY:
The study is designed to evaluate the effect of parenteral glutamine supplementation on infection in burn patients.

DETAILED DESCRIPTION:
Despite improvements in prevention and management, burn injury continues to represent a major threat to the health and welfare of people worldwide in all age groups. Even with early surgical intervention and aggressive antibiotic therapy, infectious complications are a major cause of death in severe burn injury, accounting for 75% of all deaths occurring after initial resuscitation.

It is proposed that one source of these infections is a translocation of gram-negative bacteria from the gut. However, this mechanism of bacterial translocation through the gut wall remains a controversial mechanism of infection in humans. In animal studies, it has been demonstrated that glutamine supplementation can decrease gut-derived bacterial translocation and improve outcomes from burn injury.

Whether this holds true in humans has to be evaluated by additional studies. A recent study concluded that glutamine supplementation reduces gram-negative bacteremia in burned patients but viewed itself as preliminary and suggested that more clinical trials are warranted to corroborate the study outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 years.
* Total burn surface area of 20% - 60%.
* Expected length of stay in ICU > 48 hr.
* Admission within 72 hrs of burn injury.
* Any thermal injury such as flame burns. Scald burns and contact burns.

Exclusion Criteria:

* Burn patients with hepatic failure.
* Burn patient with Severe renal failure (glomerular filtration rate (eGFR <50 ml/min).
* Patients with inborn errors of amino-acid metabolism (e.g., phenylketonuria).
* Burn patients with pre-existing severe cardiac, pulmonary diseases.
* Burn patients with diabetes mellitus or cancer.
* Patients with metabolic acidosis (pH<7.35).
* Electric burns.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
wound culture test | on 1,5,10 and 15 days after ICU admission
  whether +ve or -ve test

SECONDARY OUTCOMES:
Procalcitonin level | on 1,5,10 and 15 days after ICU admission
  ng/ml
CRP | on 1,5,10 and 15 days after ICU admission
  mg/litre

CONTACTS AND LOCATIONS:
Locations (1):
- Ashraf Magdy Eskandr, Shibeen Elkoom, Egypt

IPD SHARING:
Plan to Share IPD: No
Data will be available with after the end of the study when requested